CLINICAL TRIAL: NCT00509691
Title: A Phase I Trial to Examine the Safety, Clinical, Immunologic and Virologic Effects of CMV pp65 Specific Cytotoxic T Lymphocytes for Recipients of Allogeneic Stem Cell Transplants With Persistent or Therapy Refractory Infections
Brief Title: Vaccine Therapy in Treating Patients Who Have Undergone a Donor Stem Cell Transplant and Have Cytomegalovirus Infection That Has Not Responded to Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000557037; PSCI-25114
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: infection; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; high risk metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent breast cancer; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; recurrent Wilms tumor and other childhood kidney tumors; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma; stage IIA ovarian epithelial cancer; stage IIA ovarian germ cell tumor; stage IIB ovarian epithelial cancer; stage IIB ovarian germ cell tumor; stage IIC ovarian epithelial cancer; stage IIC ovarian germ cell tumor; stage IIIA ovarian epithelial cancer; stage IIIA ovarian germ cell tumor; stage IIIB ovarian epithelial cancer; stage IIIB ovarian germ cell tumor; stage IIIC ovarian epithelial cancer; stage IIIC ovarian germ cell tumor; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Neoplasms; Infections; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Breast Neoplasms; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Wilms Tumor; Leukemia, Hairy Cell; Multiple Myeloma | interventions — Polymerase Chain Reaction; Flow Cytometry; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental)
  Interventions: Biological: cytomegalovirus pp65-specific cytotoxic T lymphocytes; Genetic: polymerase chain reaction; Other: diagnostic laboratory biomarker analysis; Other: flow cytometry; Other: immunologic technique

INTERVENTIONS:
Biological: cytomegalovirus pp65-specific cytotoxic T lymphocytes
Genetic: polymerase chain reaction
Other: diagnostic laboratory biomarker analysis
Other: flow cytometry
Other: immunologic technique

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill cytomegalovirus infections.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients who have undergone a donor stem cell transplant and have cytomegalovirus infection that has not responded to therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety of infusing cytomegalovirus (CMV) pp65-specific cytotoxic T-lymphocytes (CTL) generated using pp65 peptides in patients who have undergone allogeneic stem cell transplantation and have persistent CMV infections.

Secondary

* Characterize CMV pp65-specific immune responses in terms of cytotoxicity and cytokine production pre-infusion and then periodically thereafter.
* Characterize the levels of CMV DNA in recipients of CMV pp65 CTL and observe whether the CTL infusion has any impact on the level of virus.

OUTLINE: This is a multicenter study.

Patients receive cytomegalovirus (CMV) pp65 cytotoxic T-cell infusion on day 1. Patients may receive up to 2 more doses at least 2 weeks after previous dose.

Blood samples are collected and analyzed by quantitative CMV PCR, chromium release assays for CMV pp65-specific cytotoxicity, and immunophenotype for CD3, CD4, CD8, CD56, CD19, and CD45 RA/RD. Intracellular cytofluorometry is used to assess IL-2, IL-4, IL-10, and IFN-γ production by CD4 and CD8 CMV-specific effector cells.

After completion of study treatment, patients are followed periodically for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytomegalovirus (CMV) seropositive

  * Patient has had CMV antigenemia for ≥ 2 weeks OR CMV DNA levels ≥ 600 copies/μg of DNA despite antiviral therapy targeting CMV (ganciclovir or foscarnet)
* No prior allogeneic stem cell transplantation before the most recent transplantation
* CMV seropositive donor negative for HIV-1, HIV-2, HTLV-1/2 available

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2 (for patients ≤ 16 years of age) OR Lansky performance status 70-100%
* Bilirubin < 2.0 mg/dL
* AST and ALT < 2.5 times upper limit of normal
* Creatinine clearance > 50 mL/min
* Pulse oximetry > 95% without supplemental oxygen
* No history of graft-vs-host disease (GVHD) ≥ grade 2
* Not moribund
* No patients not expected to survive 1 month after T cell infusion due to cardiac, pulmonary, renal, hepatic, or neurologic dysfunction

PRIOR CONCURRENT THERAPY:

* No concurrent systemic immunosuppressive agents for the treatment of GVHD

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Toxicity | 1 year
Treatment failure | 1 year
Safety | 1 year

SECONDARY OUTCOMES:
Time to development of cytomegalovirus (CMV) specific immune reconstitution | 1 year
CMV DNA levels | 1 year
Time during post-infusion follow up at which the dominant CMV pp65 epitope for the donor is recognized by the cytotoxic t-cell lymphocyte recipient | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States